CLINICAL TRIAL: NCT02731105
Title: Pilot Study of Tolerability and Effectivity Following Application of Two Combination Topical Acne Products Clindamycin 1% and 0.025% Tretinoin Gel (Acnatac® Gel), Adapalen 0,1% and Benzoyl Peroxide 2,5% Gel (Epiduo® Gel)
Brief Title: Pilot Study of Tolerability and Effectivity of Two Combination Topical Acne Products
Acronym: PREFECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GWT-TUD GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PREFECT-trial
Record Dates: First submitted 2016-03-29; First posted 2016-04-07 (Estimated); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Acne Vulgaris
Keywords: acne; vulgaris; Clindamycin; Tretinoin; Adapalen; Benzoylperoxid; Epiduo; Acnatac
MeSH Terms: conditions — Acne Vulgaris | interventions — Clindamycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Acnatac® Gel on left face and Epiduo® Gel on right face once daily for three weeks
  Interventions: Drug: Acnatac® Gel left face; Drug: Epiduo® Gel right face
- Arm 2 (Active Comparator): Epiduo® Gel on left face and Acnatac® Gel on right face once daily for three weeks
  Interventions: Drug: Acnatac® Gel right face; Drug: Epiduo® Gel left face

INTERVENTIONS:
Drug: Acnatac® Gel left face — topical application
  Other Names: Clindamycin 1%, Tretinoin 0,025%
  Arms: Arm 1
Drug: Epiduo® Gel right face — topical application
  Other Names: Adapalen 0,1% and Benzoylperoxid 2,5%
  Arms: Arm 1
Drug: Acnatac® Gel right face — topical application
  Other Names: Clindamycin 1%, Tretinoin 0,025%
  Arms: Arm 2
Drug: Epiduo® Gel left face — topical application
  Other Names: Adapalen 0,1% and Benzoylperoxid 2,5%
  Arms: Arm 2

SUMMARY:
Study to compare two gels that are used to treat acne vulgaris. It will be compared the tolerability and effectivity following application of two combination topical acne products clindamycin 1% and 0.025% tretinoin gel (Acnatac® Gel), adapalen 0,1% and benzoyl peroxide 2,5% gel (Epiduo® Gel).

DETAILED DESCRIPTION:
At baseline, data will be collected regarding demographics and medical/medication histories, lesions will be counted and a medical examination will be done. Female patients who could be pregnant will be tested by using a pregnancy test. Each patient receives two tubes with different medication that has to be applied on the left or right side of their face each by themselves at home once a day(Acnatac® Gel, Duac® Gel, Epiduo® Gel).

Patients and study-center staff will be instructed not to reveal the treatment allocation to the investigator, and patients will be instructed not to apply the product in their presence Follow-up visits will be conducted on days 0, 7 and 21. On these days the investigator measures erythema and dryness/scaling using the Investigators´Global Assessment, the severity of burning/ stinging and itching by using Study Subject Self-Assessment, records the number of acneiform lesions, measures health-related quality of life using DLQI-Score, skin hydration using Corneometer, transepidermal water loss (TEWL) using Tewameter®, skin surface pH using pH-Meter and skin sebum excretion using Sebumeter.

On days 0, 7, and 21 it will be collected information about current use of any other medication. Adverse events (AEs) and serious adverse events (SAEs) will be monitored at each visit. On day 21 there will be made a last pregnancy test. Checking compliance will be made regularly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of mild to moderate facial acne vulgaris at baseline
* Age: 14 years to 50 years
* No evidence of facial irritation (erythema, dryness/scaling, burning/itching/stinging) that is not typical for acne vulgaris
* Willingness to take part in acne study including screening visit and follow up visits on day 0,7, and 21
* No use of systemic antibiotics, steroids, retinoids and keratolytics within the last 30 days before start of the acne study
* Patients have to sign personally consent form and follow study procedures
* Patient is in good general health

Exclusion Criteria:

* Female patients who were pregnant, planning to become pregnant or breastfeeding
* Sexually active female subjects do not use a medically acceptable form of contraception (oral contraception, injectable or implantable methods or intrauterine devices)
* Female patients who are in childbearing years except post-menopausal (12 month natural amenorrhoea),

  ▪ postoperative (6 weeks after ovariectomy with or without hysterectomy)
* regularly and correct use of contraceptive with error rate < 1 %/year
* no sex
* vasectomy of the partner
* Diseases of the facial skin other than acne
* No concomitant topical medications (including make-up) or keratolytics as sulphur, salicylic acid, benzoyl peroxide, resorcin and abradents and acid-containing peels one week before the study starts
* Patients who had facial procedures (chemical peel, laser therapy, photodynamic therapy, microdermabrasion, or UV light therapy) within the past 4 weeks
* No concomitant participation in other studies within the past 30 days
* Hypersensitivity against any ingredients of Acnatac® -gel or Epiduo®gel
* Systemic medication with antibiotics or antibiotics within the last 4 weeks before study start
* Systemic medication with retinoids within the last 6 months before study start
* Topical treatment of acne vulgaris within the last two weeks before study
* Acne fulminans,
* Severe systemic disease respectively taking immunosuppressive drugs
* Severe liver disease
* Severe renal disease
* History or presence of regional enteritis or inflammatory bowel disease
* Other reasons that the doctor in charge decides about

Ages: 14 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2015-02; Primary Completion 2017-02-21 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
transepidermal water loss (TEWL) | 3 weeks

SECONDARY OUTCOMES:
Measuring the severity of burning/ stinging and itching using Study Subject Self-Assessment | 3 weeks
Measuring and recording the number of acneiform lesions | 3 weeks
Measuring health-related quality of life using DLQI-Score/CDLQI | 3 weeks
Measuring skin surface pH using pH-Meter | 3 weeks
Measuring skin sebum excretion using Sebumeter | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Roland Aschoff, MD, Principal Investigator — Uniklinikum Dresden
Locations (1):
- Universitätsklinikum Carl Gustav Carus; Klinik und Poliklinik für Dermatologie, Dresden, Saxony, Germany